CLINICAL TRIAL: NCT02664194
Title: Hypothermia as an Adjunctive Therapy to Percutaneous Intervention in Patients With Acute Myocardial Infarction
Acronym: COOL-MI InCor
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sao Paulo General Hospital (Other)
Collaborators: ZOLL Circulation, Inc., USA (Industry)
Responsible Party: Principal Investigator, Luís Augusto Palma Dallan, MD, University of Sao Paulo General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16568; 0242/11 (Other: Cappesq); 3575/10/164 (Other: Sdc)
Record Dates: First submitted 2016-01-18; First posted 2016-01-26 (Estimated); Last update posted 2018-05-11 (Actual); Status verified 2018-05

CONDITIONS: Hypothermia, Induced; Rewarming; Myocardial Infarction; Percutaneous Cornonary Intervention
Keywords: Hypothermia; Rewarming; Myocardial Infarction; Percutaneous Cornonary Intervention
MeSH Terms: conditions — Hypothermia; Myocardial Infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Control Group (Active Comparator): Primary percutaneous coronary intervention only
  Interventions: Procedure: Primary Percutaneous Coronary Intervention
- 03 Hours Hypothermia Group - Proteus® Cooling System (Experimental): 03 hours of intravascular hypothermia as an adjunctive method to primary percutaneous coronary intervention, adjunct hypothermia methods and parameters using Proteus® Cooling System.
  Interventions: Device: Proteus® Cooling System; Procedure: Primary Percutaneous Coronary Intervention
- 01 Hour Hypothermia Group - Proteus® Cooling System (Experimental): 01 hour of intravascular hypothermia as an adjunctive method to primary percutaneous coronary intervention, adjunct hypothermia methods and parameters using Proteus® Cooling System.
  Interventions: Device: Proteus® Cooling System; Procedure: Primary Percutaneous Coronary Intervention

INTERVENTIONS:
Device: Proteus® Cooling System — Intravascular hypothermia as an adjunctive method to primary percutaneous coronary intervention, adjunct hypothermia methods and parameters, using Proteus® Cooling System.
  Other Names: Cooling / Hypothermia
  Arms: 01 Hour Hypothermia Group - Proteus® Cooling System; 03 Hours Hypothermia Group - Proteus® Cooling System
Procedure: Primary Percutaneous Coronary Intervention — Primary percutaneous coronary intervention
  Other Names: Primary Angioplasty

SUMMARY:
To evaluate and improve the safety and efficacy of hypothermia as an adjunctive therapy to percutaneous coronary intervention in patients with acute myocardial infarction.

DETAILED DESCRIPTION:
Single-center, prospective, randomized, controlled clinical study involving at least 70 patients with up to 10 roll-in patients (for training purposes).

Male and female adults presenting with acute myocardial infarction may be eligible for this research study. To qualify, patients must go to the Emergency Room within up to 6 hours of onset of chest pain, present with anterior or inferior acute myocardial infarction with elevation of the ST segment greater than 1mm in 2 or more contiguous leads in the anterior or inferior wall and be eligible for the performance of a percutaneous intervention procedure.

The intervention will be intravascular hypothermia using Proteus System® as an adjunctive method to percutaneous coronary intervention, adjunct hypothermia methods and parameters.

During the randomization phase, at least 70 patients who meet the eligibility criteria will be randomly assigned to the 03 hour hypothermia group (percutaneous coronary intervention + cooling), to the 01 hour hypothermia group (percutaneous coronary intervention + cooling) or to the control group (percutaneous coronary intervention only) in a 1:1:1 ratio.

All patients receiving PCI + Cooling will also be randomized to groups A and B. Group A will receive 1 liter of chilled normal saline (4°C) prior to PCI/reperfusion, and Group B will not receive chilled normal saline (4°C), prior to PCI.

All patients included in the randomization phase will be included in the statistical analysis.

Approximately 10 Roll-in patients may be enrolled at the center (for training purpose), with anterior or inferior wall infarcts.

The primary endpoint will be reduction of the infarct size (%LV), studied with cardiac magnetic resonance imaging (cMR) using late gadolinium enhancement 5 days after the AMI, and 30 days after the infarction.

The secundary endpoints will be

* incidence of major adverse cardiac events (MACE) or death within 30 days;
* resolution of the ST segment elevation after PCI;
* ejection fraction determined by cMR after 30 days.
* evaluation of adverse events potentially related to hypothermia and/or endovascular cooling within 30 days.
* Differences in plaquelet aggregation during cooling and rewarming.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged > 18 years.
* The patient must have symptoms consistent with an acute myocardial infarction (chest pain, that is, pain in the arm, etc.) that do not improve with nitroglycerin, with an onset of symptoms greater than 30 minutes but less than six hours before admission to the emergency room.
* Roll-In Patients: Anterior or Inferior MI with ST-segment elevation of > 1mm in two or more contiguous anterior precordial or inferior leads.
* Randomized Patients: Anterior wall AMI with elevation of ST segment > 1mm in two or more anterior precordial contiguous leads.
* Patient must be eligible for PCI.
* The patient or the patient's legal guardian agrees to and is willing to sign the informed consent form to participate in the clinical study (for countries where appropriate).

Exclusion Criteria:

* The patient had a previous myocardial infarction.
* The patient is experiencing cardiogenic shock (systolic blood pressure (SBP) < 80 mmHg and not responsive to fluids, or SBP < 100 mmHg with vasopressors, or in need of an intra-aortic balloon - IAB).
* The patient is presenting with resuscitated cardiac arrest, atrial fibrillation or Killip risk Stratification class II through IV.
* The patient has aortic dissection or requires an immediate surgical or procedural intervention other than PCI.
* The patient has known Congestive Heart Failure (CHF), hepatic failure, end-stage kidney disease or sever renal failure (clearance < 30 ml/min/1.73m2 .
* The patient is febrile (temperature > 37.5 °) or has experienced an infection with fever in the last 5 days.
* The patient has known previous CABG.
* The patient has known recent stroke within 90 days of admission.
* Cardiopulmonsary decompensation that has occurred en route to the hospital or in the opinion of the physician that is imminent or likely to occur following presentation to the clinical site.
* Contraindications to hypothermia, such as patients with known hematologic dyscrasias which affect thrombosis 9e.g., cryoglobulinemia, sickle cell disease, serum cold agglutinins) or vasospastic disorders (such as Raynaud's or thromboangitis obliterans.
* The patient has a known hypersensitivity or contraindication to aspirin, heparin, or sensitivity to contrast [agents], which cannot be adequately pre-medicated.
* The patient has a known history of bleeding diathesis, coagulopathy, cryoglobulinemia or sickle cell anemia, or will refuse blood transfusion.
* The patient is < 1.5 m (4 feet 11 inches) tall.
* The patient has a known hypersensitivity to buspirone hydrochloride or meperidine and/or was treated with a monoamine oxidase inhibitor in the last 14 days.
* The patient has a known history of severe hepatic or renal failure, untreated hypothyroidism, Addison's disease, benign prostatic hypertrophy or urethral stricture, that in the opinion of the physician, would be incompatible with the administration of pethidine/meperidine.
* The patient has an Inferior Vena Cava filter in place (IVC).
* The patient has a pre-MI life expectancy < 1 year due to underlying medical conditions or pre-existing morbidities.
* The patient has a known, unresolved history of drug use or alcohol dependency, or is not able to comprehend or follow the instructions.
* The patient is currently enrolled in another investigational drug or device trial that has not completed the primary endpoint. (Note: For the purpose of this protocol, patients involved in extended follow-up trials for products that were investigational but are currently commercially available are not considered enrolled in an investigational trial).
* The patient is apprehensive about or unwilling to undergo the required MRI imaging at follow-up, has a documented or suspected diagnosis of claustrophobia, or has Gadolinium allergy, or is in permanent Atrial Fibrillation.
* The patient has received thrombolytic therapy en route to the hospital
* The patient shows clinical evidence of spontaneous reperfusion as observed symptomatically and/ or from ECG findings (partial or complete ST resolution in ECG before randomization) upon admission
* The patient is a vulnerable subject, for instance, a person in detention (i.e., prisoner or ward of the state)
* The patient is a female who is known to be pregnant.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2016-01; Primary Completion 2019-01 (Estimated); Study Completion 2019-07 (Estimated)

PRIMARY OUTCOMES:
Infarct size | 30 days after STEMI
  Reduction of the infarct size (%LV), studied with cardiac magnetic resonance imaging(cMR) using late gadolinium enhancement 5 days after the AMI, and 30 days after the infarction.
Ejection fraction | 30 days after STEMI
  ejection fraction (%) as determined cardiac resonance imaging (cMR) at 30 days after randomization.
MACE | 30 days after STEMI
  Incidence up to 30 days after randomization of major adverse cardiac events (MACE), defined as: death related to cardiac complications, recurrent AMI or need for revascularization of the target vessel.

SECONDARY OUTCOMES:
ST Segment Elevation | 3 hours after STEMI
  Resolution of the ST segment elevation (milimiters) after PCI.
Cardiac enzymes | 30 days after STEMI
  Serial evaluation of cardiac enzymes (Troponin I - ng/mL) in order to provide a secondary measure of cell injury
Composite of adverse events | 30 days after STEMI
  Composite of adverse events, defined as:
  1. All-cause mortality
  2. Recurrent AMI
  3. Need for revascularization of the target vessel
  4. Cerebral vascular accident
  5. Cardiogenic shock
  6. Pulmonary embolism
  7. Ventricular fibrillation
  8. Vascular complications requiring surgery
  9. Bleeding requiring transfusion of 2 or more units of red blood cell concentrate
Device complications | 30 days after STEMI
  Complications potentially related to the implantation or to the use of the ZOLL System (hematoma, venous puncture, vascular complications requiring surgery, bleeding, surgical wound infection, systemic infection, deep venous thrombosis, pulmonary embolism by tomography)
Cooling complications | 30 days after STEMI
  Potential complications related to cooling (thermal discomfort, myocardial ischemia, coagulopathy, arrhythmias, hypotension and pulmonary edema).
All cause mortality | 30 days after STEMI
  All cause mortality
Anterior MI | 30 days after STEMI
  Patients with elevation of the ST segment greater than 1mm in 2 or more contiguous leads in the anterior wall (v1 to v6)
03 hours versus 01 hour cooling | 30 days after STEMI
  Comparison of three hours of cooling versus one hour of cooling regarding infarct size (%LV) as determined by study with cardiac magnetic resonance

CONTACTS AND LOCATIONS:
Overall Officials: Sergio Timerman, PhD, Principal Investigator — InCor - FMUSP; Pedro A Lemos, PhD, Principal Investigator — InCor - FMUSP
Locations (1):
- InCor - Instituto do Coracao - HCFMUSP, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Dae MW, Gao DW, Ursell PC, Stillson CA, Sessler DI. Safety and efficacy of endovascular cooling and rewarming for induction and reversal of hypothermia in human-sized pigs. Stroke. 2003 Mar;34(3):734-8. doi: 10.1161/01.STR.0000057461.56040.FE. Epub 2003 Feb 13. PMID 12624300
- [Result] Gotberg M, Olivecrona GK, Koul S, Carlsson M, Engblom H, Ugander M, van der Pals J, Algotsson L, Arheden H, Erlinge D. A pilot study of rapid cooling by cold saline and endovascular cooling before reperfusion in patients with ST-elevation myocardial infarction. Circ Cardiovasc Interv. 2010 Oct;3(5):400-7. doi: 10.1161/CIRCINTERVENTIONS.110.957902. Epub 2010 Aug 24. PMID 20736446
- [Derived] Dallan LAP, Dae M, Giannetti NS, Polastri TF, Lima MKF, Rochitte CE, Hajjar LA, San Martin CYB, Lima FG, Nicolau JC, de Oliveira MT Jr, Dallan LAO, Ribeiro da Silva EE, Kalil Filho R, Abizaid A, Lemos Neto PA, Timerman S. Endovascular therapeutic hypothermia adjunctive to percutaneous coronary intervention in acute myocardial infarction: realistic simulation as a game changer. Rev Cardiovasc Med. 2022 Mar 16;23(3):104. doi: 10.31083/j.rcm2303104. PMID 35345271
- [Derived] Dallan LAP, Giannetti NS, Rochitte CE, Polastri TF, San Martin CYB, Hajjar LA, Lima FG, Nicolau JC, Oliveira MT , Jr, Dae M, Ribeiro da Silva EE, Kalil Filho R, Lemos Neto PA, Timerman S. Cooling as an Adjunctive Therapy to Percutaneous Intervention in Acute Myocardial Infarction: COOL-MI InCor Trial. Ther Hypothermia Temp Manag. 2021 Sep;11(3):135-144. doi: 10.1089/ther.2020.0018. Epub 2020 Jun 17. PMID 32552523